CLINICAL TRIAL: NCT00193336
Title: Phase II Trial of Single Agent ZD1839 (Iressa) in Poor Performance Status Patients With Previously Untreated Advanced Non-Small Cell Lung Cancer
Brief Title: Iressa in Poor Performance Status Patients With Previously Untreated Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: SCRI Oncology Research Consortium, SCRI
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 71; IRUSIRES0002
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Lung Cancer
Keywords: NSCLC Lung Cancer; Non Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

INTERVENTIONS:
Drug: ZD1839

SUMMARY:
Because of the demonstrated single agent activity and excellent tolerability in patients with refractory non-small cell lung cancer, ZD1839 may be of benefit in the first-line treatment of patients with advanced non-small cell lung cancer who have poor performance status. In this phase II trial, we will investigate the single agent activity of first-line ZD1839 in patients with advanced non-small cell lung cancer with poor performance status

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be receive:

* ZD1839

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Biopsy proven non-small cell lung cancer
* Recurrent non-small cell lung cancer after previous surgery or radiation
* Advanced disease (stage IIIb or IV)
* No previous chemotherapy or biological therapy
* Require significant assistance with activities of daily living
* Measurable disease
* Adequate bone marrow, liver and kidney function
* Give written informed consent

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Brain metastasis
* Meningeal metastasis
* Other uncontrolled malignancies
* Women pregnant or lactating
* No measurable disease outside previous radiation therapy field

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-03; Primary Completion 2004-03 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Overall response rate

SECONDARY OUTCOMES:
Overall toxicity
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC

REFERENCES:
- [Result] Spigel DR, Hainsworth JD, Burkett ER, Burris HA, Yardley DA, Thomas M, Jones SF, Dickson NR, Scullin DC, Bradof JE, Rubinsak JR, Brierre JE, Greco FA. Single-agent gefitinib in patients with untreated advanced non-small-cell lung cancer and poor performance status: a Minnie Pearl Cancer Research Network Phase II Trial. Clin Lung Cancer. 2005 Sep;7(2):127-32. doi: 10.3816/CLC.2005.n.028. PMID 16179100
- See also: Published article in Clinical Lung Cancer — http://cigjournals.metapress.com/content/6822553744n47577/?p=0e5ad5d17e5c4241b3e7674ea8cf3df0&pi=7